CLINICAL TRIAL: NCT02846636
Title: Prospective, Multicentric, Non-controlled, Non-randomized Clinical Survey to Evaluate Mpact Cup Performance After Total Hip Arthroplasty
Brief Title: Mpact Cup Performance After Total Hip Arthroplasty
Status: Suspended | Type: Observational
Why Stopped: Surgeon stopped
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.014.07
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Total Hip Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study is to evaluate the 10 year performances of Mpact cup in total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring a total hip replacement who meets the standard indications for use for Medacta implants
* patients who accept to participate in the study
* patients who signed the consent form for the treatment of personal data

Exclusion Criteria:

* patients presenting conditions identified as contraindication for Medacta implants
* revision surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for total hip arthroplasty who meet the inclusion criteria will be invited in the study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
implant survival trough Kaplan-Meier curve | 10 years

SECONDARY OUTCOMES:
hip function with Harris Hip Score | preop, 3/6 months, 1, 3, 5, 7, 10 years
record of adverse events | intraop, 3/6 months, 1, 3, 5, 7, 10 years
implant stability trough assessment of presence of radiolucencies | 3/6 months, 1, 3, 5, 7, 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Médico-Chirurgicale Paris V, Paris, France, France

IPD SHARING:
Plan to Share IPD: No